CLINICAL TRIAL: NCT04196595
Title: Apple Women's Health Study
Status: Recruiting | Type: Observational
Sponsor: Apple Inc. (Industry)
Collaborators: Harvard School of Public Health (HSPH) (Other); National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00037562
Record Dates: First submitted 2019-11-13; First posted 2019-12-12 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Menstrual Cycle; Ovulation; Menstruation; Polycystic Ovary Syndrome; Infertility; Menopause; Reproduction; Reproductive Health
Keywords: Menstruation; Menstrual Cycle; Ovulation; Polycystic Ovary Syndrome; Infertility; Menopause; Reproduction; Reproductive Health
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational longitudinal study to advance the understanding of menstrual cycle and gynecologic health conditions including PCOS, infertility and breast cancer.The study will be hosted within the Research app(available on App Store), which allows a user to find, enroll, and participate in Apple-supported health-related research studies.

ELIGIBILITY:
Inclusion Criteria:

* Have menstruated at least once
* Be at least 18 years old (at least 19 years old in Alabama and Nebraska, at least 21 years old in Puerto Rico)
* Live in the United States of America
* Be comfortable communicating in written and spoken English
* Have installed the Apple Research app on your iPhone
* Not share your iCloud account or iPhone with anyone else
* Be willing and able to provide informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience sampling of individuals who have ever menstruated and meet other eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2019-11-14 (Actual); Primary Completion 2029-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Identify Menstrual Cycle Patterns | Up to 10 years
  Characterized using duration of menstrual flow, and cycle length in unit of days.
Epidemiologic Description of Menstrual Cycle | Up to 10 years
  Characterized using cycle patterns and self-reported demographics, no unit of measure

SECONDARY OUTCOMES:
Determine prevalence of gynecologic health conditions | Up to 10 years
  Characterized using menstrual cycle patterns and self-reported health conditions, no unit of measure

CONTACTS AND LOCATIONS:
Overall Officials: Michelle A Williams, SM, ScD, Principal Investigator — Harvard School of Public Health (HSPH); Russ B Hauser, MD, MPH, ScD, Principal Investigator — Harvard School of Public Health (HSPH); Brent A Coull, PhD, Principal Investigator — Harvard School of Public Health (HSPH); Shruthi Mahalingaiah, MD, MS, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard T.H. Chan School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhang CY, Li H, Zhang S, Suharwardy S, Chaturvedi U, Fischer-Colbrie T, Maratta LA, Onnela JP, Coull BA, Hauser R, Williams MA, Baird DD, Jukic AMZ, Mahalingaiah S, Curry CL. Abnormal uterine bleeding patterns determined through menstrual tracking among participants in the Apple Women's Health Study. Am J Obstet Gynecol. 2023 Feb;228(2):213.e1-213.e22. doi: 10.1016/j.ajog.2022.10.029. Epub 2022 Oct 29. PMID 36414993